CLINICAL TRIAL: NCT05797220
Title: Retrospective Analysis on the Efficacy of Botulinum Toxin Alone Versus Combined Botulinum Toxin and Topical Diltiazem in Chronic Anal Fissure: Short and Long-term Outcomes From a Single Center
Brief Title: The Efficacy of Botulinum Toxin Alone Versus Combined Botulinum Toxin and Topical Diltiazem in Chronic Anal Fissure
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Cigdem Arslan, Consultant Surgeon, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02-786
Record Dates: First submitted 2022-10-04; First posted 2023-04-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Anal Fissure Chronic
Keywords: botulinum toxin, anal fissure, diltiazem
MeSH Terms: conditions — Fissure in Ano | interventions — Botulinum Toxins, Type A; Diltiazem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Botulinum toxin group: The procedures were performed at outpatient clinic without anesthesia. Lyophilized 100 IU BT Type-A (BOTOX, Alergan, CA, USA) was applied after diluted with 1 cc saline. A 26-G injector was used to inject 25 unit toxin in every 4 quadrants, to the alignment of clock 12, 3, 6, and 9 to internal anal sphincters.
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]
- Botulinum toxin plus topical diltiazem group: The procedures were performed at outpatient clinic without anesthesia. Lyophilized 100 IU BT Type-A (BOTOX, Alergan, CA, USA) was applied after diluted with 1 cc saline. A 26-G injector was used to inject 25 unit toxin in every 4 quadrants, to the alignment of clock 12, 3, 6, and 9 to internal anal sphincters. After BT injection, topical 2% diltiazem gel was prescribed, applied 2 times per day for 10 days (2 doses of 1 gr each per day). No selection criteria were used when recommending this treatment; it was randomly suggested to some for a while during the cohort since the surgeon believed it might enhance the efficacy of BT.
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox] + Diltiazem Hydrochloride 20 Mg/G Rectal Gel

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Botox]
  Groups: Botulinum toxin group
Drug: Botulinum Toxin Type A Injection [Botox] + Diltiazem Hydrochloride 20 Mg/G Rectal Gel
  Groups: Botulinum toxin plus topical diltiazem group

SUMMARY:
Anal fissure (AF) is a painful tear extending from the anal canal to the dentate line. Although the exact pathophysiology is not known, an increase in anal tonus, decreased ano-dermal blood flow and local ischemia are possible mechanisms. The most effective treatment modality in chronic AF is lateral internal sphincterotomy however, incontinence rates are still reported as high as 8-30%. Topical diltiazem and botulinum toxin (BT) injection are good alternatives to surgery with lack of persistent side effects, easy applicability, and reproducibility, however, recurrence rates were reported up to 50% for each. A combination of BT with topical diltiazem may provide better results in terms of healing and recurrence. In this retrospective analysis a comparison of BT injection alone and BT injection combined with topical diltiazem treatment was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complaints longer than 8 weeks (chronic anal fissure)
* Patients who completed at least 24 months of follow-up (3rd day, 10th day, 1st-month, and 2nd-month face-to-face clinic visits and 6, 12, and 24 months phone calls)
* Patients who received conservative treatments including topical diltiazem and nitrites

Exclusion Criteria:

* Patients with previous anal surgery (lateral internal sphincterotomy, hemorrhoidectomy, anal fistula)
* Patients with inflammatory bowel diseases
* Patients with accompanying anorectal disease (hemorrhoids, anal fistula, abscess)
* Patients who underwent botulinum toxin injection within 1 year before recruitment
* Patients with anterior, lateral, or multiple fissures
* Comorbidities (AIDS, sexually transmitted disease, tuberculosis, leukemia)
* Pregnancy
* Prescription of calcium canal blockers or nitrites
* Hypersensitivity to diltiazem or botulinum toxin
* Patients without anal pain

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Female and males older than 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Fissure healing at 1 month | 1 month
  Evaluation of complete epithelization of the fissure by the principal investigator by rectal examination
Days to pain-free defecation | 1 month
  Patient reported time until pain-free defecation. This will be evaluated on 3rd day, 10th day and 1-month outpatient visits.

SECONDARY OUTCOMES:
Complete healing at 48 months | 48 months
  Any recurrent symptoms evaluated by the surgeon within 2 months in the outpatient clinic and reported by the patient at phone call follow-up at 6 months, 12 months, 24 months, and 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Cigdem Arslan, MD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Other (Non U.s.), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I don not have a website to share IPD however if required I can share datasets, protocols and other information.